CLINICAL TRIAL: NCT03455985
Title: Effectiveness of a Diabetes Focused Discharge Order Set Among Poorly Controlled Hospitalized Patients Transitioning to Glargine U300 Insulin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interruption of study enrollment and procedures due to COVID-19 health crisis
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kathleen Dungan, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017H0354
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2; Patient Discharge; Blood Glucose, Low; Blood Glucose, High
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Discharge Order Set (DOS) (Experimental): Patients in the DOS group will receive instructions for self-titration of basal insulin as part of the discharge order. The DOS contains a comprehensive checklist for basic diet, hospital follow-up, glucose targets and instructions for monitoring, insulin pens and pen needles, glucose testing supplies, and ancillary orders. Phone calls will assess adherence with instructions for self-titration. Glucose lowering medication management following discharge will otherwise be conducted by the patient's usual or designated standard of care provider.
  Interventions: Other: Discharge Order Set (DOS)
- Enhanced Standard Care (ESC) (Other): Patients in the ESC group will receive hospital discharge instructions using current best practices within the overall functionality of the electronic medical record, which facilitates medication reconciliation and use of a patient care resource manager. Phone calls are information gathering only in the ESC group, and questions related to care will be referred to the usual provider.
  Interventions: Other: Enhanced Standard Care (ESC)

INTERVENTIONS:
Other: Discharge Order Set (DOS) — In addition to the elements in ESC, for the DOS group the primary team will be contacted to complete the Diabetes Discharge order set, which will be pre-populated into the electronic discharge navigator. Follow-up phone calls in the DOS group will also assess and reinforce insulin dose self-titration.
  Arms: Discharge Order Set (DOS)
Other: Enhanced Standard Care (ESC) — Patients in the ESC group will receive hospital discharge instructions using current best practices within the overall functionality of the electronic medical record, which facilitates medication reconciliation and use of a patient care resource manager. Phone calls are information gathering only in the ESC group, and questions related to care will be referred to the usual provider.
  Arms: Enhanced Standard Care (ESC)

SUMMARY:
Diabetes is present in 25% of hospitalized patients; yet effective hospital discharge programs for patients with diabetes are understudied. In particular, patients who are initiating or intensifying insulin therapy have the most to benefit in terms of glycemic control. However, these patients are also particularly vulnerable to poor transitions of care for a variety of reasons, including the complexity of therapy, inadequate patient education, differences in patient and provider expectations, and insufficient resources. Disruption of insulin therapy following hospitalization is associated with higher HbA1c, shorter survival, and increased readmissions and medical costs. In a Society of Hospital Medicine Survey, only one fourth of hospitals were supported with written protocols to standardize medication, education, equipment, and follow-up instructions. However, discharge order sets have largely been limited to the inpatient setting and have not been utilized to guide insulin use at hospital discharge. This study will assess whether a nurse supported diabetes focused inpatient discharge order set (DOS) can improve post-discharge outcomes among hospitalized patients with poorly controlled insulin-requiring diabetes.

DETAILED DESCRIPTION:
In this 24 week randomized controlled trial, hospitalized insulin-requiring patients with type 2 diabetes and poor glycemic control (HbA1c >8.5%) will receive standard of care insulin therapy including basal insulin glargine U300 (TOUJEO®) plus additional background therapy (non-insulin and prandial insulin therapies) with either a diabetes focused discharge order set (DOS) and follow-up communication to facilitate insulin titration and outpatient follow-up or enhanced standard care (ESC). 222 patients (type 2 diabetes) will be recruited. Hospitalized patients with type 2 diabetes (HbA1c >8.5%) who are receiving basal insulin at least 10 unit per day and are able to provide informed consent and complete study procedures will be approached. All patients will be discharged on glargine U300 with initial doses determined by the discharging team. Patients in the DOS group will receive instructions for self-titration of basal insulin as part of the discharge order. The DOS contains a comprehensive checklist for basic diet, hospital follow-up, glucose targets and instructions for monitoring, insulin pens and pen needles, glucose testing supplies, and ancillary orders. Patients will have follow-up phone calls at week 2, 6, and in-person visits at week 12 and 24. Phone calls will assess adherence with instructions for self-titration in the DOS group but are information gathering only in the ESC group, and questions related to care will be referred to the usual provider. Glucose lowering medication management following discharge will otherwise be conducted by the patient's usual or designated standard of care provider. The study and all study-related documents will be approved by the OSU IRB. All data analyses will be completed as intention to treat analyses. Longitudinal outcomes (e.g., HbA1c) will be analyzed using mixed models utilizing all available measurements from individuals randomized.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes, type 2 ≥3 months duration
* HbA1c >8.5%
* Ages 25-75 years
* Phone or electronic media availability
* Receiving basal insulin >10 unit/day

Exclusion Criteria:

* Sensitive admissions: Prisoners
* Pregnancy
* Unable to consent or follow study directions in English
* Expected nursing facility stay longer than 2 weeks

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Dungan, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook CB, Seifert KM, Hull BP, Hovan MJ, Charles JC, Miller-Cage V, Boyle ME, Harris JK, Magallanez JM, Littman SD. Inpatient to outpatient transfer of diabetes care: planing for an effective hospital discharge. Endocr Pract. 2009 Apr;15(3):263-9. doi: 10.4158/EP.15.3.263. PMID 19364697
- [Background] Dungan K, Lyons S, Manu K, Kulkarni M, Ebrahim K, Grantier C, Harris C, Black D, Schuster D. An individualized inpatient diabetes education and hospital transition program for poorly controlled hospitalized patients with diabetes. Endocr Pract. 2014 Dec;20(12):1265-73. doi: 10.4158/EP14061.OR. PMID 25100371
- [Background] Wexler DJ, Beauharnais CC, Regan S, Nathan DM, Cagliero E, Larkin ME. Impact of inpatient diabetes management, education, and improved discharge transition on glycemic control 12 months after discharge. Diabetes Res Clin Pract. 2012 Nov;98(2):249-56. doi: 10.1016/j.diabres.2012.09.016. Epub 2012 Oct 1. PMID 23036785
- [Background] Kimmel B, Sullivan MM, Rushakoff RJ. Survey on transition from inpatient to outpatient for patients on insulin: what really goes on at home? Endocr Pract. 2010 Sep-Oct;16(5):785-91. doi: 10.4158/EP10013.OR. PMID 20350914
- [Background] Wheeler K, Crawford R, McAdams D, Robinson R, Dunbar VG, Cook CB. Inpatient to outpatient transfer of diabetes care: perceptions of barriers to postdischarge followup in urban African American patients. Ethn Dis. 2007 Spring;17(2):238-43. PMID 17682352
- [Background] Dungan KM. The effect of diabetes on hospital readmissions. J Diabetes Sci Technol. 2012 Sep 1;6(5):1045-52. doi: 10.1177/193229681200600508. PMID 23063030
- [Background] Wu EQ, Zhou S, Yu A, Lu M, Sharma H, Gill J, Graf T. Outcomes associated with insulin therapy disruption after hospital discharge among patients with type 2 diabetes mellitus who had used insulin before and during hospitalization. Endocr Pract. 2012 Sep-Oct;18(5):651-9. doi: 10.4158/EP11314.OR. PMID 22440990
- [Background] Rodriguez A, Magee M, Ramos P, Seley JJ, Nolan A, Kulasa K, Caudell KA, Lamb A, MacIndoe J, Maynard G. Best Practices for Interdisciplinary Care Management by Hospital Glycemic Teams: Results of a Society of Hospital Medicine Survey Among 19 U.S. Hospitals. Diabetes Spectr. 2014 Aug;27(3):197-206. doi: 10.2337/diaspect.27.3.197. PMID 26246780
- [Background] Wright A, Feblowitz JC, Pang JE, Carpenter JD, Krall MA, Middleton B, Sittig DF. Use of order sets in inpatient computerized provider order entry systems: a comparative analysis of usage patterns at seven sites. Int J Med Inform. 2012 Nov;81(11):733-45. doi: 10.1016/j.ijmedinf.2012.04.003. Epub 2012 Jul 18. PMID 22819199
- [Background] Neinstein A, MacMaster HW, Sullivan MM, Rushakoff R. A detailed description of the implementation of inpatient insulin orders with a commercial electronic health record system. J Diabetes Sci Technol. 2014 Jul;8(4):641-51. doi: 10.1177/1932296814536290. Epub 2014 May 25. PMID 24876450
- [Background] Yu CH, Sun XH, Nisenbaum R, Halapy H. Insulin order sets improve glycemic control and processes of care. Am J Med. 2012 Sep;125(9):922-8.e4. doi: 10.1016/j.amjmed.2012.02.018. Epub 2012 Jul 14. PMID 22800878
- [Background] Noschese M, Donihi AC, Koerbel G, Karslioglu E, Dinardo M, Curll M, Korytkowski MT. Effect of a diabetes order set on glycaemic management and control in the hospital. Qual Saf Health Care. 2008 Dec;17(6):464-8. doi: 10.1136/qshc.2006.021790. PMID 19064664
- [Background] Schnipper JL, Liang CL, Ndumele CD, Pendergrass ML. Effects of a computerized order set on the inpatient management of hyperglycemia: a cluster-randomized controlled trial. Endocr Pract. 2010 Mar-Apr;16(2):209-18. doi: 10.4158/EP09262.OR. PMID 20061280
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Barr CC. Retinopathy and nephropathy in patients with type 1 diabetes four years after a trial of intensive insulin therapy, by The Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. N. Engl. J. Med 342:381-9, 2000. Surv Ophthalmol. 2001 Mar-Apr;45(5):459-60. doi: 10.1016/s0039-6257(01)00187-4. No abstract available. PMID 11274700
- [Background] Hoerger TJ, Segel JE, Gregg EW, Saaddine JB. Is glycemic control improving in U.S. adults? Diabetes Care. 2008 Jan;31(1):81-6. doi: 10.2337/dc07-1572. Epub 2007 Oct 12. PMID 17934153
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. In 2007. Diabetes Care. 2008 Mar;31(3):596-615. doi: 10.2337/dc08-9017. PMID 18308683
- [Background] Krop JS, Powe NR, Weller WE, Shaffer TJ, Saudek CD, Anderson GF. Patterns of expenditures and use of services among older adults with diabetes. Implications for the transition to capitated managed care. Diabetes Care. 1998 May;21(5):747-52. doi: 10.2337/diacare.21.5.747. PMID 9589235
- [Background] Calver J, Brameld KJ, Preen DB, Alexia SJ, Boldy DP, McCaul KA. High-cost users of hospital beds in Western Australia: a population-based record linkage study. Med J Aust. 2006 Apr 17;184(8):393-7. doi: 10.5694/j.1326-5377.2006.tb00289.x. PMID 16618238
- [Background] Johansen H, Nair C, Bond J. Who goes to the hospital? An investigation of high users of hospital days. Health Rep. 1994;6(2):253-77. English, French. PMID 7873720
- [Background] Zook CJ, Moore FD. High-cost users of medical care. N Engl J Med. 1980 May 1;302(18):996-1002. doi: 10.1056/NEJM198005013021804. PMID 6767975
- [Background] Howell S, Coory M, Martin J, Duckett S. Using routine inpatient data to identify patients at risk of hospital readmission. BMC Health Serv Res. 2009 Jun 9;9:96. doi: 10.1186/1472-6963-9-96. PMID 19505342
- [Background] Shipton S. Risk factors associated with multiple hospital readmissions. Home Care Provid. 1996 Mar-Apr;1(2):83-5. doi: 10.1016/s1084-628x(96)90234-8. PMID 9157913
- [Background] Jacob L, Poletick EB. Systematic review: predictors of successful transition to community-based care for adults with chronic care needs. Care Manag J. 2008;9(4):154-65. doi: 10.1891/1521-0987.9.4.154. PMID 19177973
- [Background] Bersoux S, Cook CB, Kongable GL, Shu J. Trends in glycemic control over a 2-year period in 126 US hospitals. J Hosp Med. 2013 Mar;8(3):121-5. doi: 10.1002/jhm.1997. Epub 2012 Dec 19. PMID 23255411
- [Background] Shepperd S, McClaran J, Phillips CO, Lannin NA, Clemson LM, McCluskey A, Cameron ID, Barras SL. Discharge planning from hospital to home. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD000313. doi: 10.1002/14651858.CD000313.pub3. PMID 20091507
- [Background] Robbins JM, Webb DA. Diagnosing diabetes and preventing rehospitalizations: the urban diabetes study. Med Care. 2006 Mar;44(3):292-6. doi: 10.1097/01.mlr.0000199639.20342.87. PMID 16501402
- [Background] Moghissi ES, Korytkowski MT, DiNardo M, Einhorn D, Hellman R, Hirsch IB, Inzucchi SE, Ismail-Beigi F, Kirkman MS, Umpierrez GE; American Association of Clinical Endocrinologists; American Diabetes Association. American Association of Clinical Endocrinologists and American Diabetes Association consensus statement on inpatient glycemic control. Endocr Pract. 2009 May-Jun;15(4):353-69. doi: 10.4158/EP09102.RA. No abstract available. PMID 19454396
- [Background] Umpierrez GE, Reyes D, Smiley D, Hermayer K, Khan A, Olson DE, Pasquel F, Jacobs S, Newton C, Peng L, Fonseca V. Hospital discharge algorithm based on admission HbA1c for the management of patients with type 2 diabetes. Diabetes Care. 2014 Nov;37(11):2934-9. doi: 10.2337/dc14-0479. Epub 2014 Aug 28. PMID 25168125
- [Background] Varroud-Vial M. Improving diabetes management with electronic medical records. Diabetes Metab. 2011 Dec;37 Suppl 4:S48-52. doi: 10.1016/S1262-3636(11)70965-X. PMID 22208710
- [Background] Weber V, Bloom F, Pierdon S, Wood C. Employing the electronic health record to improve diabetes care: a multifaceted intervention in an integrated delivery system. J Gen Intern Med. 2008 Apr;23(4):379-82. doi: 10.1007/s11606-007-0439-2. PMID 18373133
- [Background] Schnipper JL, Hamann C, Ndumele CD, Liang CL, Carty MG, Karson AS, Bhan I, Coley CM, Poon E, Turchin A, Labonville SA, Diedrichsen EK, Lipsitz S, Broverman CA, McCarthy P, Gandhi TK. Effect of an electronic medication reconciliation application and process redesign on potential adverse drug events: a cluster-randomized trial. Arch Intern Med. 2009 Apr 27;169(8):771-80. doi: 10.1001/archinternmed.2009.51. PMID 19398689
- [Background] Moore P, Armitage G, Wright J, Dobrzanski S, Ansari N, Hammond I, Scally A. Medicines reconciliation using a shared electronic health care record. J Patient Saf. 2011 Sep;7(3):148-54. doi: 10.1097/PTS.0b013e31822c5bf9. PMID 21857238
- [Background] Kramer JS, Hopkins PJ, Rosendale JC, Garrelts JC, Hale LS, Nester TM, Cochran P, Eidem LA, Haneke RD. Implementation of an electronic system for medication reconciliation. Am J Health Syst Pharm. 2007 Feb 15;64(4):404-22. doi: 10.2146/ajhp060506. PMID 17299180
- [Background] Staroselsky M, Volk LA, Tsurikova R, Newmark LP, Lippincott M, Litvak I, Kittler A, Wang T, Wald J, Bates DW. An effort to improve electronic health record medication list accuracy between visits: patients' and physicians' response. Int J Med Inform. 2008 Mar;77(3):153-60. doi: 10.1016/j.ijmedinf.2007.03.001. Epub 2007 Apr 16. PMID 17434337
- [Background] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708
- [Background] Umpierrez GE, Hor T, Smiley D, Temponi A, Umpierrez D, Ceron M, Munoz C, Newton C, Peng L, Baldwin D. Comparison of inpatient insulin regimens with detemir plus aspart versus neutral protamine hagedorn plus regular in medical patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 Feb;94(2):564-9. doi: 10.1210/jc.2008-1441. Epub 2008 Nov 18. PMID 19017758
- [Background] Garber AJ. Will the next generation of basal insulins offer clinical advantages? Diabetes Obes Metab. 2014 Jun;16(6):483-91. doi: 10.1111/dom.12219. Epub 2013 Oct 31. PMID 24118819
- [Background] Steinstraesser A, Schmidt R, Bergmann K, Dahmen R, Becker RH. Investigational new insulin glargine 300 U/ml has the same metabolism as insulin glargine 100 U/ml. Diabetes Obes Metab. 2014 Sep;16(9):873-6. doi: 10.1111/dom.12283. Epub 2014 Mar 24. PMID 24571126
- [Background] Riddle MC, Bolli GB, Ziemen M, Muehlen-Bartmer I, Bizet F, Home PD; EDITION 1 Study Investigators. New insulin glargine 300 units/mL versus glargine 100 units/mL in people with type 2 diabetes using basal and mealtime insulin: glucose control and hypoglycemia in a 6-month randomized controlled trial (EDITION 1). Diabetes Care. 2014 Oct;37(10):2755-62. doi: 10.2337/dc14-0991. Epub 2014 Jul 30. PMID 25078900
- [Background] Yki-Jarvinen H, Bergenstal R, Ziemen M, Wardecki M, Muehlen-Bartmer I, Boelle E, Riddle MC; EDITION 2 Study Investigators. New insulin glargine 300 units/mL versus glargine 100 units/mL in people with type 2 diabetes using oral agents and basal insulin: glucose control and hypoglycemia in a 6-month randomized controlled trial (EDITION 2). Diabetes Care. 2014 Dec;37(12):3235-43. doi: 10.2337/dc14-0990. Epub 2014 Sep 5. PMID 25193531
- [Background] Bolli GB, Riddle MC, Bergenstal RM, Ziemen M, Sestakauskas K, Goyeau H, Home PD; on behalf of the EDITION 3 study investigators. New insulin glargine 300 U/ml compared with glargine 100 U/ml in insulin-naive people with type 2 diabetes on oral glucose-lowering drugs: a randomized controlled trial (EDITION 3). Diabetes Obes Metab. 2015 Apr;17(4):386-94. doi: 10.1111/dom.12438. Epub 2015 Feb 12. PMID 25641260
- [Background] Ritzel R, Roussel R, Bolli GB, Vinet L, Brulle-Wohlhueter C, Glezer S, Yki-Jarvinen H. Patient-level meta-analysis of the EDITION 1, 2 and 3 studies: glycaemic control and hypoglycaemia with new insulin glargine 300 U/ml versus glargine 100 U/ml in people with type 2 diabetes. Diabetes Obes Metab. 2015 Sep;17(9):859-67. doi: 10.1111/dom.12485. Epub 2015 Jun 16. PMID 25929311
- [Background] Healy SJ, Black D, Harris C, Lorenz A, Dungan KM. Inpatient diabetes education is associated with less frequent hospital readmission among patients with poor glycemic control. Diabetes Care. 2013 Oct;36(10):2960-7. doi: 10.2337/dc13-0108. Epub 2013 Jul 8. PMID 23835695
- [Background] Mistry R, Rosansky J, McGuire J, McDermott C, Jarvik L; UPBEAT Collaborative Group. Social isolation predicts re-hospitalization in a group of older American veterans enrolled in the UPBEAT Program. Unified Psychogeriatric Biopsychosocial Evaluation and Treatment. Int J Geriatr Psychiatry. 2001 Oct;16(10):950-9. doi: 10.1002/gps.447. PMID 11607938
- [Background] Anderson ES, Winett RA, Wojcik JR. Self-regulation, self-efficacy, outcome expectations, and social support: social cognitive theory and nutrition behavior. Ann Behav Med. 2007 Nov-Dec;34(3):304-12. doi: 10.1007/BF02874555. PMID 18020940
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Mitchell SE, Sadikova E, Jack BW, Paasche-Orlow MK. Health literacy and 30-day postdischarge hospital utilization. J Health Commun. 2012;17 Suppl 3:325-38. doi: 10.1080/10810730.2012.715233. PMID 23030580
- [Background] Weiss BD, Mays MZ, Martz W, Castro KM, DeWalt DA, Pignone MP, Mockbee J, Hale FA. Quick assessment of literacy in primary care: the newest vital sign. Ann Fam Med. 2005 Nov-Dec;3(6):514-22. doi: 10.1370/afm.405. PMID 16338915
- [Background] Anderson RM, Fitzgerald JT, Gruppen LD, Funnell MM, Oh MS. The Diabetes Empowerment Scale-Short Form (DES-SF). Diabetes Care. 2003 May;26(5):1641-2. doi: 10.2337/diacare.26.5.1641-a. No abstract available. PMID 12716841
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Oakes JM, Feldman HA. Statistical power for nonequivalent pretest-posttest designs. The impact of change-score versus ANCOVA models. Eval Rev. 2001 Feb;25(1):3-28. doi: 10.1177/0193841X0102500101. PMID 11205523
- [Background] International Hypoglycaemia Study Group. Erratum to: Glucose concentrations of less than 3.0 mmol/l (54 mg/dl) should be reported in clinical trials: a joint position statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetologia. 2017 Feb;60(2):377. doi: 10.1007/s00125-016-4168-0. No abstract available. PMID 27921135
- [Background] Mehrotra DV, Li X, Liu J, Lu K. Analysis of longitudinal clinical trials with missing data using multiple imputation in conjunction with robust regression. Biometrics. 2012 Dec;68(4):1250-9. doi: 10.1111/j.1541-0420.2012.01780.x. Epub 2012 Sep 20. PMID 22994905
- [Derived] White A, Buschur E, Harris C, Pennell ML, Soliman A, Wyne K, Dungan KM. Influence of Literacy, Self-Efficacy, and Social Support on Diabetes-Related Outcomes Following Hospital Discharge. Diabetes Metab Syndr Obes. 2022 Aug 4;15:2323-2334. doi: 10.2147/DMSO.S327158. eCollection 2022. PMID 35958875
- [Derived] White A, Bradley D, Buschur E, Harris C, LaFleur J, Pennell M, Soliman A, Wyne K, Dungan K. Effectiveness of a Diabetes-Focused Electronic Discharge Order Set and Postdischarge Nursing Support Among Poorly Controlled Hospitalized Patients: Randomized Controlled Trial. JMIR Diabetes. 2022 Jul 26;7(3):e33401. doi: 10.2196/33401. PMID 35881437
- See also: Healthcare Cost and Utilization Project. Economic and Health Costs of Diabetes — http://archive.ahrq.gov/data/hcup/highlight1/high1.pdf
- See also: Toujeo prescribing instructions — http://products.sanofi.us/toujeo/toujeo.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Discharge Order Set (DOS) | Enhanced Standard Care (ESC)
Started | 82 | 76
Completed | 44 | 45
Not Completed | 38 | 31

BASELINE CHARACTERISTICS:
Population: Analysis population is the same as the participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Discharge Order Set (DOS) | Enhanced Standard Care (ESC) | Total
Number analyzed (Participants) | 82 | 76 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 67 | 139
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (10.1) | 51.4 (10.5) | 51.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 35 | 33 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 80 | 75 | 155
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 41 | 41 | 82
  White | 40 | 34 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 82 | 76 | 158

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to 24 Weeks
Description: We will test for a difference in 24 week change in HbA1c between the DOS and ESC groups using a linear mixed model for the longitudinal HbA1c measurements. A Wald test of the treatment-by-time interaction will be used to test our primary hypothesis that DOS affects 24 weeks change in Hb1Ac.
Time Frame: 24 weeks
Population: Data were collected at study visits and extracted from the electronic medical records.
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Discharge Order Set (DOS) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 44 | 45
percentage of glycosylated hemoglobin | -2.1 (0.3) | -1.0 (0.3)
Statistical Analysis 1: Comparison: Discharge Order Set (DOS) vs Enhanced Standard Care (ESC); Test type: Superiority; p = 0.09, Regression, Linear; Mean Difference (Net) = 0.07, Standard Error of Mean 0.4

2. Secondary Outcome: Change in HbA1c From Baseline to 12 Weeks
Description: We will test for a difference in 24 week change in HbA1c between the DOS and ESC groups using a linear mixed model for the longitudinal HbA1c measurements. A Wald test of the treatment-by-time interaction will be used to test our primary hypothesis that DOS affects 12 weeks change in Hb1Ac.
Time Frame: 12 weeks
Population: HbA1c was obtained from study visits as well as from the electronic medical record.
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Discharge Order Set (DOS) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 54 | 54
percentage of glycosylated hemoglobin | -2.0 (0.3) | -1.4 (0.3)
Statistical Analysis 1: Comparison: Discharge Order Set (DOS) vs Enhanced Standard Care (ESC); Test type: Superiority; p = 0.20, Regression, Linear; Mean Difference (Net) = -0.5, Standard Error of Mean 0.4

3. Secondary Outcome: Proportion Using Insulin Glargine U300 at 24 Weeks
Description: proportion of patients who remain on insulin glargine U300 at 24 weeks The difference in proportions of patients who remain on insulin glargine U300 at 24 weeks between treatment groups will be computed and compared using test of proportions.
Time Frame: 24 weeks
Population: The difference in proportions of patients who remain on insulin glargine U300 at 24 weeks between treatment groups will be computed and compared using test of proportions.
Measure: Count of Participants; unit: Participants
Arm/Group | Discharge Order Set (DOS) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 32 | 30
Participants | 25 | 25
Statistical Analysis 1: Comparison: Discharge Order Set (DOS) vs Enhanced Standard Care (ESC); Test type: Superiority; p > 0.99, Fisher Exact

4. Secondary Outcome: Fasting Glucose
Description: We will test for a difference in fasting glucose between the DOS and ESC groups using a linear mixed model.
  reported measure differs from original plan due to lack of fasting glucose in hospitalized patients.
Time Frame: 24 weeks
Population: Data were collected from study visits from participants who were fasting.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Discharge Order Set (DOS) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 20 | 21
mg/dl | 152.5 [127.3 to 247.3] | 209 [129.5 to 234]
Statistical Analysis 1: Comparison: Discharge Order Set (DOS) vs Enhanced Standard Care (ESC); Test type: Superiority; p = 0.39, Regression, Linear; Mean Difference (Final Values) = -26.5, Standard Error of Mean 30.3

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events will include severe hypoglycemia rates, pregnancy, overdose, and breach of confidentiality. In addition the following definitions apply:
  DEFINITIONS
  Serious adverse event (SAE): any untoward medical occurrence including:
  * Results in death, hospitalization, disability, congenital anomaly
  * Is life threatening,
  * Is a medically important event or reaction. Related Adverse Event, i.e. Adverse Drug Reaction Unexpected Adverse Event New Safety finding
Arm/Group | Discharge Order Set (DOS) | Enhanced Standard Care (ESC)
All-Cause Mortality (participants affected / at risk) | 1/82 | 0/76
Serious Adverse Events (participants affected / at risk) | 30/82 | 34/76
Other Adverse Events (participants affected / at risk) | 0/82 | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discharge Order Set (DOS) (N=82) | Enhanced Standard Care (ESC) (N=76)
Severe hypoglycemia (Endocrine disorders) | 5 (5) | 8 (10) — hypoglycemia associated with seizure or hemodynamic compromise or in need of outside assistance
Hyperglycemia (Endocrine disorders) | 3 (3) | 2 (4)
Diabetic ketoacidosis (Endocrine disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
hyperkalemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar degenerative disc disease (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 0 (0) | 2 (2)
wound infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
foot ulcer (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
lower extremity edema (Vascular disorders) | 0 (0) | 1 (1)
arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
clostridium dificile collitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
hypertensive urgency (Cardiac disorders) | 1 (2) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
cervical stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
heart failure (Cardiac disorders) | 2 (2) | 5 (6)
dental abscess (Infections and infestations) | 0 (0) | 1 (1)
dacroadenitis (Eye disorders) | 0 (0) | 1 (1)
fall (General disorders) | 1 (1) | 0 (0)
angina (Cardiac disorders) | 1 (1) | 0 (0)
cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
hernia (Surgical and medical procedures) | 1 (1) | 0 (0)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was stopped early due to loss to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03455985/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03455985/ICF_001.pdf